CLINICAL TRIAL: NCT04479072
Title: Aspirin to Prevent Cardiac Dysfunction in Preeclampsia
Brief Title: Aspirin and Preeclampsia
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Prevention
Other Study IDs: IRB18-1606
Record Dates: First submitted 2020-07-13; First posted 2020-07-21 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: Preeclampsia Postpartum
Keywords: Preeclampsia; Postpartum GLS Levels; Postpartum Activin A Levels; Aspirin; Cardiac Postpartum Therapy; Hypertension; Cardiovascular disease
MeSH Terms: conditions — Pre-Eclampsia; Hypertension; Cardiovascular Diseases | interventions — Aspirin

STUDY DESIGN:
Intervention Model Description: Main Study: Subjects will be randomized to two arms. One arm will receive a daily dose of aspirin 81 mg, starting at their baseline visit. The other arm will receive daily dose of placebo pill at their baseline visit. There will be a third arm, where subjects will not receive any study drug and will be considered the observational arm.
  Sub-Study: Subjects who completed the main part of the study and choose to participate will be randomized once more into one of two arms for the purposes of the sub-study. One arm will receive the GDMP, which includes the RPM program. The other arm will not receive the GDMP and will continue thier usual standard of care course per thier treating physician.
Who Masked: Participant, Investigator
Masking Description: The study team and all randomized subjects will be blinded to which arm they were placed in during the main part of the study. Subjects in the observational group will not be randomized and not given an intervention.
  The sub-study portion has no blinding attached to it
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Intervention Arm (Active Comparator): 60 subjects will be randomly assigned to this arm. The subjects in this arm will receive a daily dose of aspirin 81 mg.
  Interventions: Drug: Aspirin 81 mg
- Placebo Arm (Placebo Comparator): 60 subjects will be randomly assigned to this arm. The subjects in this arm will receive a daily dose of a placebo pill
  Interventions: Drug: Placebo
- Observational Arm (No Intervention): 60 subjects will be placed in the observational arm. These subjects will not receive any intervention but will be followed and asked to return at the same time interval as the other 2 groups.

INTERVENTIONS:
Drug: Aspirin 81 mg — Subjects in the interventional arm will receive a daily dose of aspirin 81 mg, starting at their baseline visit and to be taken up to their 6-month follow-up visit.
  Other Names: acetylsalicylic acid 81 mg
  Arms: Intervention Arm
Drug: Placebo — Subjects in this group will receive a daily dose of a placebo pill, starting at their baseline visit and to be taken up to their 6-month follow-up visit.
  Arms: Placebo Arm

SUMMARY:
This is a single-center, double-blind, randomized, placebo-controlled clinical trial. Peripartum and postpartum Activin A are significantly elevated in women with preeclampsia. Our hypothesis is that elevated Activin A levels reflect a remediable signal and that reducing postpartum Activin A levels with aspirin therapy will improve (GLS) in preeclamptic patients.

DETAILED DESCRIPTION:
The primary objective of the main part of this trial is to mechanistically compare the effect of postpartum aspirin therapy versus placebo in preeclamptic patients identified as high risk for postpartum cardiac dysfunction using Activin A. The intent is to evaluate the effect of selective treatment based on Activin A status rather than treatment for all postpartum preeclamptic women.

After informed consent, 5cc of blood will be collected from the median cubital vein on antepartum admission to labor and delivery for Activin A screening. The patient will be subjected to a total of 2 such blood draws- a single draw at screening, one at their 6 month postpartum visit. The member of the study team carrying out the blood draw will immediately label the specimen in the presence of the subject, after the collection and before leaving the patient's bedside, room, cubicle or surgical suite. The guidelines from, "The University of Chicago Medicine Policy and Procedure Manual - Phlebotomy Service Infection Control 04-26" will be followed for specimen collection and transport. Activin A levels based on our previous data will be classified as elevated if greater than 23.74 ng/ml in the last trimester of pregnancy (4). This threshold was selected on the basis of our prior data suggesting an inflection point in the rate of abnormal GLS postpartum at this concentration. Patients with elevated Activin A levels will be randomized to a placebo group receiving routine postpartum cardiovascular standard of care or to an intervention arm with 81 mg daily aspirin therapy added to care at their postpartum delivery stay. The rationale for only randomizing women with elevated Activin A levels is that among women with an elevated Activin A antepartum, 85% developed abnormalities in GLS at one year postpartum versus 25% in women with non-elevated Activin A levels. Women whose Activin A levels are not elevated will receive the same care as that provided to the placebo group and will also be followed for one year (n=60). All other subjects who meet the criterial of elevated Activin A levels, will either be randomized to the aspirin therapy group (N = 60) or a placebo group (N = 60). The investigators choose postpartum Aspirin therapy post-delivery to avoid any immediate delivery or C-section associated bleeding complications and to coincide with their postpartum well-baby visit.

The investigator will determine the blood Activin A levels at 6 months after delivery, measured using ELISA. The samples will be assayed for Activin A level using commercially available ELISA kits (Ansh Labs; Webster, TX) following the manufacturer's recommendations. Each sample will be run in triplicate and the values averaged. GLS at 6 months after delivery will be measured using fully automated vendor-independent software that uses a computer learning algorithm to facilitate endocardial border detection.

Mean arterial pressure, and other indices of systolic and diastolic function (ejection fraction (EF), early filling/atrial contraction (E/A), deceleration time (DT), mitral annular motion (E'), and left atrial volume index) measured at the baseline and 6 months postpartum. Transthoracic echocardiograms will be performed and reported according to American Society of Echocardiography guidelines. Ejection fraction and left atrial volume will be calculated using the Simpson's biplane disc method. Left ventricular mass index (LVMI) will be calculated using the area length method.

ELIGIBILITY:
Inclusion Criteria:

1. Pregnant Adults between 18 and 45 years of age
2. Diagnosed with preeclampsia
3. Presenting for delivery with a singleton gestation.

Exclusion Criteria:

1. We will exclude patients in labor
2. Patients with preexisting cardiomyopathy, chronic hypertension, ischemic or valvular heart disease, pulmonary disease, diabetes mellitus, chronic kidney disease, multiple gestation
3. Plan to deliver outside of the participating site
4. Co-enrolled in other trials that might affect the patients taking the study medication, as determined by the PI.
5. Aspirin allergy
6. Clear indication for aspirin therapy or contraindication to aspirin therapy
7. Clinically significant conditions that might limit adherence to trial regimen (e.g., peptic ulcer disease, history of gastrointestinal bleeds, bleeding disorders)
8. Currently or planning on taking any nonsteroidal anti-inflammatory drugs while they are participating in this study.
9. Those who cannot provide consent

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Pregnant women with preeclampsia
Enrollment: 180 (Estimated)
Dates: Start 2021-02-15 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Difference in Activin A levels | 6 Months
  The primary outcome will compare Activin A levels at 6 months between patients randomized to aspirin therapy versus placebo and the observational group.
GLS percentages | 6 months
  The primary outcome will compare GLS levels as a percentage (%) at 6 months between patients randomized to aspirin therapy versus placebo and the observational group.

SECONDARY OUTCOMES:
Mean Arterial Pressure | 6 Months
  Difference in mean arterial pressure in subjects, from their baseline to 6 month TTE
Ejection Fraction % | 6 Months
  Comparing the difference in the ejection fraction percentages, from the subjects baseline to 6 month TEE.
Deceleration Time | 6 Months
  Comparing the difference between deceleration time from subjects from their baseline to 6 month TTE.
Mitral Annular Motion | 6 Months
  Comparing the difference between mitral annular motion, in millimeters (mm), from subjects baseline to 6 month TTE.
Left Atrial Volume Index | 6 Months
  Comparing the difference between left atrial volume index, from the subjects baseline to 6 month TTE.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Chicago Hospital, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No